CLINICAL TRIAL: NCT02167191
Title: Determining the Effectiveness of a High Intensity Interval Training Exercise Programme in the Healthy, Elderly Population
Brief Title: HIT in the Healthy Elderly Population
Acronym: HIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HIT
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Interval Training; Pre Operative Exercise; Prehabilitation; Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIT (Experimental): High intensity interval training sessions on an cycle ergometer
  Interventions: Behavioral: HIT

INTERVENTIONS:
Behavioral: HIT — 12 sessions of HIT exercise in 31 days on a stationary cycle ergometer

SUMMARY:
It is widely known that exercise improves general fitness and that fitter patients recover more easily from illness and surgery. Conversely, unfit patients have a significantly higher morbidity and mortality after surgery and a longer inpatient stay. This will become increasingly important in an aging population as baseline fitness generally declines with age.

One method of improving cardiovascular fitness is by using low intensity endurance training programmes, a disadvantage of these it that they can take several months to show improvement. High intensity interval training (HIT) programmes that use short episodes of high intensity exercise have also been shown to improve fitness. These HIT programmes have also shown improvement in functional capacity and quality of life in patients with chronic disease. An advantage of HIT is that improvements in fitness may occur in a shorter time than traditional endurance training. It is also known that HIT can give superior gains over endurance training.

The primary aim of this study is to determine whether an improvement in aerobic fitness, as judged by a 2ml/kg/min increase in VO2peak, can be achieved within 31 days via a HIT programme, in a group of healthy elderly volunteers.

As a secondary aim we will assess whether this programme would be acceptable to the group studied, through determination of subject compliance and adherence to the training programme.

ELIGIBILITY:
Inclusion Criteria:

* Good health
* Male and female
* 60 -75 years old

Exclusion Criteria:

* Uncontrolled hypertension (BP > 140/100)
* Angina
* Heart failure (NYHA class III/IV)
* Cardiac arrthymias
* Right to left cardiac shunt
* Recent cardiac event
* Previous stroke/TIA
* Aneurysm (large vessel or intracranial)
* Severe respiratory disease including pulmonary hypertension
* COPD/asthma with an FEV1 less than 1.5 l
* Inclusion into any other research study in the last three months which involved: taking a drug; being paid a disturbance allowance; having an invasive procedure or exposure to ionising radiation

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
VO2 peak | 31 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Derby, Derbyshire, United Kingdom